CLINICAL TRIAL: NCT00139334
Title: Evaluate Immunogenicity, Reactogenicity & Safety of 2 Doses of GSK Biologicals' Oral Live Attenuated HRV Vaccine (RIX4414 at 106.5 CCID50) When Given Concomitantly With OPV Versus Given Alone (HRV Vaccine Dose Given 15 Days After the OPV Dose) in Healthy Infants in Bangladesh
Brief Title: A Study to Test 2 Doses of the HRV Vaccine Given With or Without OPV in Healthy Infants in Bangladesh
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 103992; NCT00209976 (obsolete NCT alias)
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections

INTERVENTIONS:
Biological: Rotavirus

SUMMARY:
The main objective of this study is to provide immunogenicity data for GSK Biologicals' HRV vaccine when co-administered with OPV or when given alone (HRV vaccine dose given 15 days after the OPV dose).

DETAILED DESCRIPTION:
"The study will have four groups: Group HRV + OPV, Group HRV alone, Group Placebo + OPV and Group Placebo alone. Two-dose immunisation will be administered in healthy infants at approximately 12 and 16 weeks of age. Immunogenicity, reactogenicity and safety relative to the placebo will also be evaluated. Treatment allocation: randomized (2:2:1:1). Routine EPI vaccines should be administered during the study following the EPI recommendation in Bangladesh."

ELIGIBILITY:
Inclusion criteria:

* Healthy infants aged 6 weeks±1 at first study vaccination.

Exclusion criteria:

* Malnutrition, no history of rotavirus gastroenteritis, allergic disease or chronic gastrointestinal disease, not received protocol-prohibited treatment.

Ages: 5 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300
Dates: Start 2005-06; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Endpoints : Safety/immunogenicity.Immunogenicity of GSK Biologicals' HRV vaccine in terms of anti-rotavirus IgA antibody seroconversion at Visit 6 in the group receiving of HRV vaccine concomitantly with OPV versus placebo group.

SECONDARY OUTCOMES:
Immunogenicity of GSK Biologicals' HRV vaccine in terms of anti-rotavirus IgA antibody seroconversion, vaccine take, and rotavirus shedding at Visit 6 in each group; Immunogenicity of OPV at Visit 6 in each group; Reactogenicity and safety in each group.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bhattacharya SK et al. Immune response in infants sero-positive at pre-vaccination: Human rotavirus vaccine Rotarix™. Abstract presented at 5th World Congress WSPID, Bangkok, Thailand, 15-18 November 2007.
- [Background] Zaman et al. Immunogenicity of an Oral Polio Vaccine is Unaffected when Co-Administered with a Human Rotavirus Vaccine in Bangladeshi Children. Absract presented at 5th World Congress WSPID, Bangkok, Thailand, 15-18 November 2007.
- [Background] Zaman K, Sack DA, Yunus M, Arifeen SE, Podder G, Azim T, Luby S, Breiman RF, Neuzil K, Datta SK, Delem A, Suryakiran PV, Bock HL; Bangladeshi Rotavirus Vaccine study group. Successful co-administration of a human rotavirus and oral poliovirus vaccines in Bangladeshi infants in a 2-dose schedule at 12 and 16 weeks of age. Vaccine. 2009 Feb 25;27(9):1333-9. doi: 10.1016/j.vaccine.2008.12.059. Epub 2009 Jan 20. PMID 19162114
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 103992 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103992 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103992 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103992 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103992 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103992 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register